CLINICAL TRIAL: NCT05530577
Title: Effects of Semaglutide on Nicotine Intake and Smoking Lapse
Brief Title: Effects of Semaglutide on Nicotine Intake
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-1548; R21DA047663-02 (NIH)
Record Dates: First submitted 2022-08-26; First posted 2022-09-07 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Use Disorder; Nicotine Addiction
MeSH Terms: conditions — Tobacco Use Disorder | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Randomized parallel group design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide via subcutaneous injections at escalating doses (0.25mg to 1.0mg) over 9 weeks.
  Interventions: Drug: Semaglutide
- Sham/Placebo (Sham Comparator): Participants will receive sham subcutaneous injections over 9 weeks.
  Interventions: Drug: Sham/placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide (subcutaneous)
  Arms: Semaglutide
Drug: Sham/placebo — Sham subcutaneous injection
  Arms: Sham/Placebo

SUMMARY:
Tobacco use remains the foremost cause of preventable deaths in the U.S. and worldwide. Advancing new smoking cessation therapies, including those targeting novel biological mechanisms, is a critical public health priority. Accumulating evidence from preclinical studies suggests that glucagon-like peptide-1 (GLP-1) receptor agonists reduce intake and/or reinstatement of addictive drugs, including nicotine. However, translational work is necessary to establish whether GLP-1 receptor agonists alter aspects of nicotine response and smoking behavior in smokers. Human laboratory studies play a pivotal role in drug development by providing a time- and cost-efficient means of validating preclinical findings, also providing an ideal platform for studying mechanisms of medication effects. This is an experimental investigation to examine the effects of an approved GLP-1 receptor agonist on nicotine intake and reinstatement. Dependent smokers will be enrolled in a double-blind, parallel-arm trial with laboratory endpoints. Laboratory procedures will include a validated procedure for measuring smoking lapse/reinstatement after overnight abstinence. This study will provide initial laboratory evidence for the potential efficacy of GLP-1 receptor agonists as adjunctive treatments for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Smoking 5+ cigarettes per day (on average) over the past year, with no period of abstinence > 90 days
* Biochemical verification of smoking status, based on expired CO > 8 at baseline
* Willingness to take study medication and complete study procedures
* Willingness to complete lab sessions involving cigarette smoking
* Ability to communicate in English

Exclusion Criteria:

* Regular use of electronic nicotine delivery systems (ENDS/vaping), cigars, chewing tobacco or snuff, based on at least weekly use in the past 30 days
* Past 30-day use of nicotine replacement therapies/products
* Reporting past 30-day use of illicit drugs other than cannabis at baseline, or having a positive toxicology screen for illicit drugs other than cannabis at baseline
* Current engagement in alcohol or smoking cessation treatments, or currently engaged in intentional efforts to quit cigarette use
* Past 30-day use of: Sincalide, Sulfonylureas, insulin and insulin products or other medications that may interact with semaglutide, or weight control medications
* Prior use of semaglutide or other GLP-1 agonists
* Known or suspected hypersensitivity to study medication or related products
* Lifetime diagnosis of severe mental illness (including schizophrenia and bipolar disorder)
* Meeting criteria for current alcohol use disorder (AUD) or other substance use disorder (with the exception of tobacco or mild cannabis use disorder)
* History of suicide attempt, or recent (past 30 day) suicidal ideation, or psychiatric hospitalization in the last 6 months
* Current significant medical or neurological illness (based on self-report or medical record) including severe hepatic impairment or cirrhosis, impaired renal function (eGFR <50ml/min), acute or chronic pancreatitis, gastroparesis, gallbladder disease or cholelithiasis, other severe gastrointestinal disease, heart failure, coronary artery disease, stroke, seizure disorder, or other medical condition that poses a risk for the medication or alcohol administration components of the study (as determined by the MD)
* A personal or family history of medullary thyroid cancer or multiple endocrine neoplasia 2A or 2B
* Calcitonin greater than or equal to 50 ng/L
* Uncontrolled thyroid disease at screening
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g., subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* History of Type 1 or Type 2 diabetes, or HbA1c >6.5% measured at screening
* History of diabetic retinopathy, proliferative retinopathy, or maculopathy
* History of diabetic ketoacidosis
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ)
* Currently nursing, pregnant, anticipating pregnancy in the next 6 months, or not using a highly effective contraceptive method as judged by the MD, and defined as:

  1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  3. intrauterine device
  4. intrauterine hormone-releasing system
  5. bilateral tubal occlusion
  6. vasectomized partner
  7. sexual abstinence
* Elevation of serum lipase, amylase, direct (conjugated) bilirubin, or alkaline phosphatase (ALP), ALT, or AST) more than 3X the upper limit of normal on baseline bloodwork
* Baseline body mass index (BMI) <23kg/m^2
* Uncontrolled hypertension or systolic BP >180 mmHg and/or diastolic BP >105 mmHg, averaged from three measurements
* Plans for travel outside of the local area in the upcoming 12 weeks that would interfere with lab visits during the study period (or other logistic factors that would make it difficult to commit to entire duration of study)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hendershot, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other investigators upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available following publication of study manuscripts and will be available indefinitely.
Access Criteria: Reasonable request from qualified investigator.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Semaglutide | Sham/Placebo
Started | 12 | 12
Completed | 10 | 10
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Sham/Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (8.1) | 44.2 (5.6) | 43.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Nicotine Self-Administration
Description: Number of cigarettes smoked during a laboratory smoking procedure
Time Frame: Baseline (Week 0) to post-medication (Week 8)
Population: Analysis population includes participants who completed a post-treatment laboratory smoking session (n=10 semaglutide group, n=11 placebo group). Two participants in the semaglutide group and one participant in the placebo group discontinued participation prior to the post-treatment smoking session.
Measure: Mean (Standard Deviation); unit: Number of cigarettes
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 10 | 11
Number of cigarettes | -0.8 (0.63) | -0.5 (0.69)

2. Primary Outcome: Change in Nicotine Reinstatement Duration
Description: Duration (minutes) of resistance to smoking reinstatement during a laboratory lapse task
Time Frame: Baseline (Week 0) to post-medication (Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 10 | 11
Minutes | 10.3 (27.6) | -2.2 (20.1)

3. Secondary Outcome: Change in Daily Cigarette Smoking
Description: Number of cigarettes consumed per day during medication exposure
Time Frame: Baseline (Week 0) to study endpoint (Week 10)
Measure: Mean (Standard Deviation); unit: Number of cigarettes per day
Arm/Group | Semaglutide | Sham/Placebo
Number analyzed (Participants) | 10 | 10
Number of cigarettes per day | -3.35 (5.25) | -2.27 (4.15)

4. Other Pre Specified Outcome: Change in Cigarette Craving
Description: Self-reported craving during a cue exposure task
Time Frame: baseline (Week 0) to post-medication (Week 8)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Subjective Responses to Cigarette Smoking
Description: Self-reported responses to cigarette smoking during a laboratory smoking procedure The Cigarette Purchase Task is a 21-question self-reported measure to understand motivation for obtaining cigarettes which asks participants about the number of cigarettes they would purchase and smoke based on an increasing cigarette cost.
Time Frame: baseline (Week 0) to post-medication (Week 8)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Body Weight
Description: Body weight
Time Frame: baseline (Week 0) to study endpoint (Week 10)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in HbA1c
Description: Hemoglobin A1C (HbA1c)
Time Frame: baseline (Week 0) to study endpoint (Week 10)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the Baseline medical visit through follow-up, a total of up to 12 weeks.
Arm/Group | Semaglutide | Sham/Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Semaglutide (N=12) | Sham/Placebo (N=12)
Abdominal Pain (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 9 | 5
Vomiting (Gastrointestinal disorders) | 3 | 2
Decreased Appetite (Nervous system disorders) | 10 | 3
Fatigue (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 5 | 0
Increased Appetite (Nervous system disorders) | 0 | 2
Insomnia (Nervous system disorders) | 1 | 2
Nervousness/Anxiety (Nervous system disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT05530577/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT05530577/ICF_000.pdf